CLINICAL TRIAL: NCT03797872
Title: Clinical Effectiveness of Symptomatic Therapy Compared to Standard Step up Care for the Treatment of Low Impact Psoriatic Oligoarthritis: a 2 Arm Parallel Group Feasibility Study
Brief Title: Psoriatic Oligoarthritis Intervention With Symptomatic thErapy
Acronym: POISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/SC/0261
Record Dates: First submitted 2018-12-18; First posted 2019-01-09 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2020-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate; Sulfasalazine; Leflunomide; Methylprednisolone; Methylprednisolone Acetate; Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded assessor will perform clinical evaluations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard care (Active Comparator): Control 'step-up' therapy in the cohort (MONITOR-PsA study). Therapy for the cohort is defined by standard NHS practice. Commonly Initial therapy will be with methotrexate alone unless this is contraindicated. In cases of non-response or intolerance to methotrexate, participants will have an alternative DMARD (sulfasalazine or leflunomide). In cases of failure of two DMARDs, treatment can be escalated to biologic therapy as per National Institute for Health and Clinical Excellence (NICE) recommendations. If the requisite disease activity is not met or if there are contraindications to biologics, alternative DMARD combinations will be used.
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Leflunomide
- Local/IM steroid injections (Experimental): Symptomatic therapy arm. The intervention will delay standard treatment with disease-modifying anti-rheumatic drugs (DMARDs) and use local injections of methylprednisolone or triamcinolone to affected joints instead. Oral non-steroidal anti-inflammatory drugs (NSAIDs) will also be allowed as concomitant medication. All active joints will be treated with injections. Injections can be either be given as an intra-articular injection or as an intra-muscular injection. If any joint requires more than 2 local injections of glucocorticoid within a 6 month period, then the patient is deemed to have failed symptomatic therapy and will be withdrawn from the treatment protocol and be treated as per usual care (in most cases with DMARD therapy).
  Interventions: Drug: Methylprednisolone; Drug: Triamcinolone

INTERVENTIONS:
Drug: Methotrexate — Methotrexate up to 25mg/week as tolerated po or sc
  Other Names: methotrexate sodium
  Arms: Standard care
Drug: Sulfasalazine — Sulfasalazine up to 3g daily po
  Other Names: sulfasalazine pill
  Arms: Standard care
Drug: Leflunomide — Leflunomide 10-20mg daily po
  Other Names: leflunomide pill
  Arms: Standard care
Drug: Methylprednisolone — For IA or IM injection 20-120mg
  Other Names: methylprednisolone acetate
  Arms: Local/IM steroid injections
Drug: Triamcinolone — For IA or IM injection 20-120mg
  Other Names: triamcinolone acetonide
  Arms: Local/IM steroid injections

SUMMARY:
POISE is a two arm interventional trial nested within a cohort (Trials Within Cohorts or TWiCs design). This tests less aggressive early therapy in patients newly diagnosed with low impact oligoarticular PsA. Arm 1 will receive standard step up therapy in the cohort and act as the control group. Arm 2 will receive local steroid injections to active joints and will be able to use non-steroidal anti-inflammatory drugs (NSAIDs) only

DETAILED DESCRIPTION:
Arm 1: Control 'step-up' therapy in the cohort (MONITOR-PsA study). Therapy for the cohort is defined by standard practice in these PsA clinics following current international recommendations and National requirements for the prescription of biologic therapy. Whilst physician discretion is used, most commonly Initial therapy will be with methotrexate alone (15mg/week rising to 25mg/week as tolerated by week 8 of therapy) unless this is contraindicated. In cases of non-response or intolerance to methotrexate, participants will have an alternative DMARD (most commonly sulfasalazine or leflunomide) added or switched to at the discretion of the rheumatologist. In cases of failure of two DMARDs, treatment can be escalated to biologic therapy as per National Institute for Health and Clinical Excellence (NICE) recommendations usually with a TNF inhibitor as first line. If the requisite disease activity is not met or if there are contraindications to biologics, alternative DMARD combinations will be used. Further details are available in the PsA clinic treatment protocol which is Appendix D in the MONITOR-PsA protocol.

Arm 2: Symptomatic therapy arm. The intervention will delay standard treatment with disease-modifying anti-rheumatic drugs (DMARDs) and use local glucocorticoid injections to affected joints instead. Oral non-steroidal anti-inflammatory drugs (NSAIDs) will also be allowed as concomitant medication as indicated for individuals. Local glucocorticoid injections will include injections with methylprednisolone or triamcinolone. All active joints will be treated with glucocorticoid injections. Glucocorticoid injections can be either be given as an intra-articular injection to an inflamed joint or as an intra-muscular injection if multiple joints are involved. If any joint requires more than 2 local injections of glucocorticoid within a 6 month period, then the patient is deemed to have failed symptomatic therapy and will be withdrawn from the treatment protocol and be treated as per usual care (in most cases with DMARD therapy). If Participants require DMARD therapy, they will be offered rescue therapy as per usual clinical care but will be asked to continue with data collection for the trial. This is to ensure that sufficient data is collected for the trial but risks in delaying treatment to the individual are mitigated.

ELIGIBILITY:
Inclusion Criteria:

* Participants consented to the PsA inception cohort (MONITOR-PsA) and to be approached for alternate interventional therapies.
* Participants with mild disease as defined by:

  * Oligoarticular disease with <5 active joints at baseline assessment.
  * Low disease activity as defined by a PsA disease activity score (PASDAS) ≤3.2.
  * Low impact of disease as defined a PsA impact of disease (PSAID) ≤4.
* Participant is willing and able to give informed consent for participation in the trial.
* Male or female.
* Aged 18 years or above.
* Female Participants of child bearing potential and male Participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception (defined as true abstinence, oral contraceptives, implants, intrauterine device, barrier method with spermicide, or surgical sterilization) during the trial and for 3 months thereafter if receiving DMARD therapy (excluding sulfasalazine).
* Participant has clinically acceptable laboratory results within 6 weeks of enrolment:

  * Haemoglobin count > 8.5 g/dL
  * White blood count (WBC) > 3.5 x 109/L
  * Absolute neutrophil count (ANC) > 1.5 x 109/L
  * Platelet count > 100 x 109/L
  * ALT and alkaline phosphatase levels <3 x upper limit of normal
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her GP and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* ≥1 poor prognostic factors for psoriatic arthritis, from

  * raised C reactive protein (CRP) defined as > 4g/dl for standard non-hsCRP
  * radiographic damage defined as the presence of ≥ 1 erosion on plain radiographs of the hands and feet
  * health assessment questionnaire (HAQ) score > 1
* Contraindications to non-steroidal anti-inflammatory drugs
* Previous treatment for articular disease with synthetic DMARDs (including methotrexate, leflunomide or sulfasalazine) or biologic DMARDs (including TNF, IL12/23 or IL17 inhibitor therapies) or targeted synthetic DMARDs (PDE4 of JAK inhibitor therapies).
* Female patient who is pregnant, breast feeding or planning pregnancy during the course of the trial.
* Significant renal or hepatic impairment.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the patients at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Patients who have participated in another research trial involving an investigational product in the past 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Derived] Rombach I, Tucker L, Tillett W, Jadon D, Watson M, Francis A, Sinomati Y, Dutton SJ, Coates LC. Clinical effectiveness of symptomatic therapy compared with standard step-up care for the treatment of low-impact psoriatic oligoarthritis: the two-arm parallel group randomised POISE feasibility study. Ther Adv Musculoskelet Dis. 2022 Jan 10;13:1759720X211057668. doi: 10.1177/1759720X211057668. eCollection 2021. PMID 35035537

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The POISE trial opened on 17 April 2019 in Oxford and 19 September 2019 in Bath.
  The study remained open until 16 July 2020 as planned.
Period: Overall Study
Arm/Group | Standard Care | Local/IM Steroid Injections
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only one participant was included
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Local/IM Steroid Injections | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Are Eligible, Consent, and Complete the 48 Weeks Study
Description: To establish acceptability of this treatment approach assessing proportion of patients who are eligible, consent and complete the 48 week study. We will examine how many patients in the MONITOR cohort are eligible per year. All eligible patients in the MONITOR cohort will be approached and invited to join the study. We will then review how many patients complete the 48 week study period attending all visits from baseline to 48 weeks (0, 12, 24, 36 and 48).
Time Frame: 48 weeks
Population: All participants included
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Local/IM Steroid Injections
Number analyzed (Participants) | 1 | 0
Participants | 0 |

2. Secondary Outcome: Psoriatic Arthritis Disease Activity Score (PASDAS)
Description: A composite measure of PsA disease activity. This score is a composite measure of disease activity in PsA. There is only one total score which ranges from 0-10 with higher numbers indicating more active disease. Low disease activity is defined as <3.2.
Time Frame: 48 weeks
Population: Only one patient was recruited and he was lost to follow up before 48 weeks thus these data are not available for analysis
Arm/Group | Standard Care | Local/IM Steroid Injections
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Ultrasound Score of Synovitis
Description: A summary score of synovitis measured at baseline. The score will comprise of 23 joints bilaterally. Grey scale synovitis is scored at each site 0-3 and power doppler is also scored 0-3 at each site where higher scores indicate more severe disease. These scores are then summed to give a final score. Score range is 0-276
Time Frame: 0 weeks
Population: as for outcome 2
Arm/Group | Standard Care | Local/IM Steroid Injections
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Ultrasound Score of Enthesitis
Description: A summary score of enthesitis measured at baseline. The score will comprise of 5 entheses bilaterally. Power doppler is scored 0-3 at each site where higher scores indicate more severe disease activity. Calcifications, enthesophytes and grey scale abnormalities will each be score 0 (absent) or 1 (present) at each site. These scores are then summed to give a final score. Score range is 0-30
Time Frame: 0 weeks
Population: Only one patient was recruited and he was lost to follow up before 48 weeks thus these data are not available for analysis. The US was not performed as this was only for participants in the intervention group.
Arm/Group | Standard Care | Local/IM Steroid Injections
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 48 week study
Description: 48 week study
Arm/Group | Standard Care | Local/IM Steroid Injections
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Only 1 participants was eligible and participated in the trial during the recruitment period and this patient was lost to follow up after the baseline visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT03797872/Prot_SAP_000.pdf